CLINICAL TRIAL: NCT00479661
Title: A Prospective, Multi-centre, Randomised, Double-blind Comparison of Intravenous Dexmedetomidine With Propofol for Continuous Sedation of Ventilated Patients in Intensive Care Unit
Brief Title: Dexmedetomidine Versus Propofol for Continuous Sedation in the Intensive Care Unit (ICU)
Acronym: Prodex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Kati Kaijasilta, Orion corporation, Orion Pharma, Clinical R&D
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3005012; EudraCT 2006-006030-17
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Continuous Sedation in Initially Sedated Adults in ICU
Keywords: initial sedation; mechanical ventilation
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- 2 (Active Comparator): Propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Continuous infusion
  Arms: 1
Drug: Propofol — Continuous infusion
  Arms: 2

SUMMARY:
Patients in the ICU who need help with their breathing are put onto a machine called a ventilator and are also given a medicine, called a sedative, which helps them to sleep and makes them more comfortable. Propofol is a sedative that is routinely used for these purposes.

For most patients the aim of sedation is to make them sleepy but still able to respond to nursing staff (light sedation).

Dexmedetomidine is a new sedative for use in intensive care and in this clinical study,dexmedetomidine is compared to propofol. It is thought that dexmedetomidine might be slightly better at allowing patients to be sleepy but still respond to people around them. It also does not appear to affect patient's breathing. The purpose of this study is to test whether dexmedetomidine really does have these advantages compared to propofol.

In this study, we hope to show that: dexmedetomidine is at least as good as propofol in helping patients to sleep better and making them more comfortable, and that they are able to communicate and cooperate better with the staff treating them, and that patients treated with dexmedetomidine require a shorter time on the ventilator than those treated with propofol.

DETAILED DESCRIPTION:
This is a phase III, multi-centre, prospective, randomised, double-blind, double-dummy, active comparator study. The study consists of three periods: screening, double-dummy treatment and follow-up period.

All patients admitted to ICU will be pre-screened according to inclusion and exclusion criteria prior to informed consent using available clinical data.

Informed consent, screening and randomisation procedures should be completed within 72 hours from the time of admission to ICU and within 48 hours from starting continuous sedation. Eligible study subjects requiring light to moderate sedation (Richmond Agitation-Sedation Scale [RASS] = 0 to -3) will be randomised to either continue on propofol or switch to dexmedetomidine. Patients should not have received any other continuously or regularly administered sedative agent than propofol during the last 12 hours except for opioid analgesics. Study treatments will be titrated to achieve an individually targeted sedation range determined on a daily basis. Rescue treatment (i.e. midazolam boli) may be given if needed to achieve the target depth of sedation. Continued need for sedation will be assessed at a daily sedation stop, conducted at the same time each day. First sedation stop may be 12-36 hours from randomisation, depending on the time of day the study subject is randomised. The duration of study treatment is limited to a maximum of 14 days from randomisation. Following withdrawal of sedation, study subjects will be monitored for 48 hours and contacted by telephone 31 and 45 days after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Clinical need for sedation of an initially intubated (or tracheotomised) and ventilated (with inspiratory assistance) patient
* Prescribed light to moderate sedation (target RASS = 0 to -3) using propofol
* Patients should be randomised within 72 hours from ICU admission and within 48 hours of commencing continuous sedation in the ICU
* Patients should have an expected requirement for sedation more than 24 hours from time of randomisation
* Written informed consent must be obtained according to local regulations before starting any study procedures other than pre-screening

Exclusion Criteria:

* Acute severe intracranial or spinal neurological disorder due to vascular causes, infection, intracranial expansion or injury
* Uncompensated acute circulatory failure at time of randomisation (severe hypotension with mean arterial pressure [MAP] < 55 mmHg despite volume and pressors)
* Severe bradycardia (heart rate [HR] < 50 beats/min)
* AV-conduction block II-III (unless pacemaker installed)
* Severe hepatic impairment (bilirubin > 101 µmol/l)
* Need for muscle relaxation at the time of randomisation (may only be used for intubation and initial stabilization)
* Loss of hearing or vision, or any other condition which would significantly interfere with the collection of study data
* Burn injuries requiring regular anaesthesia or surgery
* Use of centrally acting α2 agonists or antagonists at the time of randomisation, notably clonidine
* Patients who have or are expected to have treatment withdrawn or withheld due to poor prognosis
* Patients receiving sedation for therapeutic indications rather than to tolerate the ventilator (e.g. epilepsy)
* Patients who are unlikely to require continuous sedation during mechanical ventilation (e.g. Guillain-Barré syndrome)
* Patients who are unlikely to be weaned from mechanical ventilation e.g. diseases/injuries primarily affecting the neuromuscular function of the respiratory apparatus such as clearly irreversible disease requiring prolonged ventilatory support (e.g. high spinal cord injury or advanced amyotrophic lateral sclerosis)
* Distal paraplegia
* Positive pregnancy test or currently lactating
* Received any investigational drug within the preceding 30 days
* Concurrent participation in any other interventional study (any study in which patients are allocated to different treatment groups and/or non-routine diagnostic or monitoring procedures are performed)
* Previous participation in this study
* Any other condition which, in the investigator's opinion, would make it detrimental for the subject to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Depth of sedation using the RASS. The target RASS range (target depth of sedation) should be 0 to -3 for a patient to be included in the study. The target may be amended during the study treatment, if clinically required. | 2 hourly and before each rescue treatment dose during the treatment period and the 48-hour follow-up
Duration of mechanical ventilation | Start and stop times of mechanical ventilation while the patient is treated in the ICU

SECONDARY OUTCOMES:
Nurse's assessment of subject communication with visual analogue scales (VAS) | At the end of each nursing shift during study treatment and 48 h follow-up period in the ICU
Length of ICU stay | Admission and discharge dates and times during the current ICU treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Esko Ruokonen, MD, Principal Investigator — Kuopio University Hospital; Kati Kaijasilta, MSc (Pharm), Study Director — Orion Corporation, Orion Pharma
Locations (40):
- Belgium (2):
  - Onze-Lieve-Vrouw Ziekenhuis, Anesthesia and Intensive Care Dept. Moorselbaan 164, Aalst
  - Ziekenhuis Oost-Limburg Location Sint-Jan, Dept.of Anesthesiology, Schiepse Bos, Genk
- Finland (8):
  - HUCH, Jorvi Hospital, Turuntie 150,, Espoo
  - HUCH, Meilahti Hospital, Haartmaninkatu 4, P.O.Box 340,, Helsinki
  - North Carelia Central Hospital, Tikkamaentie 16,, Joensuu
  - Kuopio University Hospital, Kuopio
  - Paijat-Hame Central Hospital, Keskussairaalankatu 7,, Lahti
  - South Carelia Central Hospital, Valto Kakelan katu 1,, Lappeenranta
  - Seinajoki Central Hospital, Hanneksenrinne 7,, Seinäjoki
  - Tampere University Hospital, ICU, Teiskonntie 35, P.O.Box 2000,, Tampere
- Germany (12):
  - Charite Berlin Klinik fur Anasthesiologie und Operative Intensivmedizin (CCM), Luisenstrasse 65 (LU 65),, Berlin
  - Universitatsklinikum Bonn, Klinik u. Poliklinik f. Anasthesiologie u., Bonn
  - Universitatsklinikum, Krankenhausstrsse 12,, Erlangen
  - Klinikum der Johann-Wolfgang-Goethe Universitat, Klinik fur Anasthesiologie,, Frankfurt am Main
  - Univ. Giessen und Marburg Abt. Anaesthesiologie, Intensivmedizin, Schmerztherapie & Palliativmedizin, Rudolf-Buchheim-Strasse 7,, Giessen
  - Universitatsklinikum Halle, Universitatsklinik fur Anasthelsiologie und Operative Intensivmedizin, Ernst-Grube Strasse 40, Halle
  - Universitatsklinikum Heidelberg Klinik fur Anasthesiologie, Im Neuenheimer Feld 110,, Heidelberg
  - Klinik fur Anasthesiologie, Intensivmedizin und Schmerztherapie, Universitatsklinikum des Saarlandes, Gebaude 57,, Homburg
  - Universitatsklinikum Leipzig, Klinik und Poliklinik fur Anaesthesiologie und Intensivtherapie, Liebigstrasse 29, Leipzig
  - Klinikum St. Georg, Delitzscher Strasse 141, Hause 20, 1. Etage, Zimmer 204, Leipzig
  - Universitatsklinikum Tubingen, Klinik fur Anasthesiologie und Intensivmedizin, Tübingen
  - Klinikum-Wetzlar-Braunfels, Forsthaus Strasse 1-3a, Wetzlar
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, Postbus 90153,, 's-Hertogenbosch
  - Westfries Gasthuis, Department Intensieve Zorgen, Maelsonstraat 3,, Hoorn
  - Rivierenland Hospital, Pres. Kennedylaan 1,, Tiel
- Russia (7):
  - Kemerovo Stte Medical Academy, 22/A Voroshilov Street, Kemerovo
  - Municipal Hospital #2, Krasnodar Diversified Treatment and Diagnostic Association, 6, Ulica Krasnykh Partizan Building 2,, Krasnodar
  - Federal State Institution Russian Centre of Functional Surgical Gastroenterology, Krasnodor Municipal Hospital, 4, ulica Sedina,, Krasnodar
  - State Institution B.B. Petrovsky Russian Research Centre of Surgery of RAMS, 2, Abrikosovsky per., Moscow
  - State Healthcare Institution V.A. Baranov Republican Hospital, 3, Pirogova Ulica,, Petrozavodsk
  - Medical Academy of Postgraduate Study, 41, ulica Kirochnaya,, Saint Petersburg
  - Federal State Healthcare Institution L.G. Sokolov Clinical Hospital, #122 of FMBA of Russia, 4, pr-t Kultury, Saint Petersburg
- Inselspital, Freiburgstsrasse 4,, Bern, Switzerland
- United Kingdom (7):
  - West Suffolk Hospital NHS Trust, Hardwick Lane, Suffolk,, Bury St Edmunds
  - Edinburgh University, Little France Crescent, Edinburgh Royal Infirmary,, Edinburgh
  - Leeds General Infirmary, Great George Street, Leeds
  - Saint John's Hospital, Howden Road West,, Livingston
  - Saint Thomas Hospital, Lambeth Palace Road,, London
  - Saint George's Hospital, Blackshaw Road, Tooting, London
  - Freeman Hospital, Freeman Road High Heaton,Newcastle Upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Turunen H, Jakob SM, Ruokonen E, Kaukonen KM, Sarapohja T, Apajasalo M, Takala J. Dexmedetomidine versus standard care sedation with propofol or midazolam in intensive care: an economic evaluation. Crit Care. 2015 Feb 19;19(1):67. doi: 10.1186/s13054-015-0787-y. PMID 25887576
- [Derived] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955